CLINICAL TRIAL: NCT04006002
Title: A Pilot Study to Compare Anatomic, Physiologic, Metabolic and Weight Changes After Standard of Care Endoscopic Gastric Restrictive Bariatric Interventions vs. Standard of Care Laparoscopic Sleeve Gastrectomy
Brief Title: Mechanism of Weight Loss After Endoscopic and Laparoscopic Sleeve Procedures
Status: Terminated | Type: Observational
Why Stopped: Not able to recruit enough patients
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Other Study IDs: 19-0112
Record Dates: First submitted 2019-06-07; First posted 2019-07-02 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-01

CONDITIONS: Weight Loss; Reflux
MeSH Terms: conditions — Weight Loss; Gastroesophageal Reflux | interventions — Metabolic Networks and Pathways

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Endoscopic Sleeve Gastrectomy: This group includes all patient who undergo Endoscopic Sleeve Gastrectomy for weight loss
  Interventions: Other: Metabolic and Hormonal profile
- Laproscopic Sleeve Gastrectomy: This group includes all patient who undergo Laproscopic Sleeve Gastrectomy for weight loss
  Interventions: Other: Metabolic and Hormonal profile

INTERVENTIONS:
Other: Metabolic and Hormonal profile — To assess changes in metabolic profiles and body metrics such as weight and BMI in these patients after an endoscopic or surgical bariatric intervention

SUMMARY:
The purpose of this research study is to understand the mechanism of weight loss for weight loss procedures: that is Laparoscopic sleeve gastrectomy and Endoscopic sleeve Gastroplasty.

DETAILED DESCRIPTION:
We want to better understand the mechanisms for weight loss by understanding the anatomic and physiologic changes that occur with gastric restrictive procedures for weight loss and to determine the differences in metabolic profile between the two restrictive procedures. We also want to identify the rate of Gastro Esophageal Reflux Disease (GERD) in patients undergoing gastric restrictive procedures for weight loss.

ELIGIBILITY:
Inclusion Criteria:

1. BMI ≥ 30 Kg/m2 scheduled to undergo a bariatric intervention
2. Patients who will be undergoing ESG or LSG as part of their clinical care Age between 18 and 75 years.
3. Both male and female subjects will be included in the study.
4. Subjects from any ethnic background will be included in the study.
5. Female participants of childbearing age should not be pregnant. (Pregnancy test will be performed on all women of child bearing potential before any standard of care endoscopic procedure. For the purpose of the study we will record that information in the patient study records).
6. Successfully complete the screening process.
7. Patients able to provide written informed consent on the IRB/EC-approved informed consent form.
8. Demonstrate willingness to follow protocol requirements, including follow-up schedule, and completion of questionnaires.
9. Having standard of care therapy (endoscopic or laproscopic) for treatment of Obesity.

Exclusion Criteria:

1. Pregnant or planning to become pregnant during period of study participation.
2. Female participants who are breast-feeding.
3. Severe Immunodeficiency.
4. Severe malnutrition.
5. The participant has life expectancy of less than 1 year due to other medical conditions.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Only participants who meet all eligibility criteria will be enrolled in the study. Participants who meet all eligibility criteria and have successfully completed the screening requirements will be asked to sign a Study Consent.
  Patients undergoing endoscopic or laparoscopic weight loss procedures will be included.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2022-01-28 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with GERD before and after intervention | 1 years
  Percentage of participants with GERD (>6% abnormal esophageal acid exposure calculated via BRAVO pH monitoring for 96 hrs ) before and at 12 months after an endoscopic or surgical bariatric intervention

SECONDARY OUTCOMES:
Compare gastric emptying after intervention | 1 year
  To compare gastric emptying and small bowel transit times, before and at 12 months after an endoscopic or surgical bariatric intervention using wireless capsule technology

CONTACTS AND LOCATIONS:
Overall Officials: Petros Benias, MD, Principal Investigator — Northwell Health
Locations (1):
- Northwell Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jirapinyo P, Thompson CC. Endoscopic Bariatric and Metabolic Therapies: Surgical Analogues and Mechanisms of Action. Clin Gastroenterol Hepatol. 2017 May;15(5):619-630. doi: 10.1016/j.cgh.2016.10.021. Epub 2016 Oct 28. PMID 27989851
- [Background] Novikov AA, Afaneh C, Saumoy M, Parra V, Shukla A, Dakin GF, Pomp A, Dawod E, Shah S, Aronne LJ, Sharaiha RZ. Endoscopic Sleeve Gastroplasty, Laparoscopic Sleeve Gastrectomy, and Laparoscopic Band for Weight Loss: How Do They Compare? J Gastrointest Surg. 2018 Feb;22(2):267-273. doi: 10.1007/s11605-017-3615-7. Epub 2017 Nov 6. PMID 29110192
- [Background] Fogel R, De Fogel J, Bonilla Y, De La Fuente R. Clinical experience of transoral suturing for an endoluminal vertical gastroplasty: 1-year follow-up in 64 patients. Gastrointest Endosc. 2008 Jul;68(1):51-8. doi: 10.1016/j.gie.2007.10.061. Epub 2008 Mar 19. PMID 18355825